CLINICAL TRIAL: NCT03909048
Title: Chronic Low Back Pain Graded - Exposure Psychoeducation Intervention
Acronym: VRGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Zina Trost, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300002878
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Pain; Low Back Pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant, statistician, and outcomes assessor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Psycho-education (Experimental): Interactive psycho-education using interactive dashboard.
  Interventions: Behavioral: Interactive - Psychoeducation
- Psycho-education (Placebo Comparator): Non-interactive psycho-education not using interactive dashboard.
  Interventions: Behavioral: Non-interactive Psychoeducation

INTERVENTIONS:
Behavioral: Interactive - Psychoeducation — Individuals will receive interactive psychoeducation in the lab over the course of a week period. Each session will take approximately 30 minutes.
  Arms: Interactive Psycho-education
Behavioral: Non-interactive Psychoeducation — Individuals will receive non-interactive psychoeducation over the course of a week period. Each session will take approximately 30 minutes.
  Arms: Psycho-education

SUMMARY:
This study will examine the effectiveness of one of two psychoeducation treatments on chronic low back pain.

DETAILED DESCRIPTION:
This study will examine the effectiveness of one of two psychoeducation treatments on chronic low back pain. Participants will be randomized to one of these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* report having low back pain for more than three months and at least half the days in the past 6 months
* be 18-65 years of age,
* have scores higher than 37 on the Tampa Scale of Kinesiophobia,

Exclusion Criteria:

* medical conditions other than back pain that significantly impair movement (e.g., arthritis)
* confirmed/suspected pregnancy
* pending litigation related to an episode of low back pain
* significant impairment in vision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity as assessed by Numeric Rating Scale | Baseline - Final assessment (average 1 week post treatment)
  The Numeric Rating Scale (NRS) measures pain intensity measured via 0-10 numeric rating scale.
  0 = No Pain - 10 = Worst Possible Pain Range of scores: 0-10
Present Pain Intensity | Baseline - Final assessment (average 1 week post treatment)
  Present Pain Intensity (PPI) assesses present pain intensity on a scale of 0 (no pain) to 5 (excruciating)
Present Pain Rating | Baseline - Final assessment (average 1 week post treatment)
  Pain Rating Index (PRI) is assessed by 15 questions assessing pain in the sensory and affective dimensions.
  Items rate from 0 (none) to 3 (severe) on degree to which the words apply to pain.
  Score Range: 0-45
Pain Chronicity assessed by the Graded Chronic Pain Scale | Baseline - Final assessment (average 1 week post treatment)
  Pain Chronicity is assessed by the Graded Chronic Pain Scale (GCPS). The GCPS is 7 questions with 3 sub-scales (Characteristic pain intensity, disability score, and disability points).
  Scoring:
  Characteristic Pain Intensity: is a 0 to 100 score derived from Questions 1 through 3: Mean (Pain Right Now, Worst Pain, Average Pain) X 10.
  Disability Score: is 0 to 100 score derived from Questions 4 through 6: Mean (Daily Activities, Social Activities, Work Activities) X 10 Disability Points: Add the indicated points for Disability Days (Question 7) and for Disability Score (0-6).
  Items rate from 0 to 10 with 0 referencing no pain/interference/change and 10 referencing pain as bad as could be/unable to carry out any activities/extreme change.
Daily Pain Monitoring: 10 point scale | Baseline - Final assessment (average 1 week post treatment)
  Daily pain monitoring defined as daily pain intensity and daily pain interference monitoring is two questions asked daily on a 10 point scale assessing daily pain and how much pain had interfered with day to day activities.
  Pain: Over the past 24 hours, how would you rate your back pain on average? (0=No Pain; 10=Worst Imaginable Pain)
  Interference: Over the past 24 hours, how much did pain interfere with your day-to-day activities? (0=No Interference; 10 = A great deal of interference)"

SECONDARY OUTCOMES:
Back Disability as assessed by the Roland Morris Disability Questionnaire | Baseline - Final assessment (average 1 week post treatment)
  The Roland Morris Disability Questionnaire (RMDQ) assesses disability due to low back pain.
  The RMDQ is a 24 item survey with yes/no response options. Score 0 -24 with ower scores indicate more impairment.
Depressive symptoms as assessed by the Center for Epidemiologic Studies Depression Scale | Baseline - Final assessment (average 1 week post treatment)
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20 item survey tool. The items are a 4 pt Likert response items.
  Scores range from 0-60 with higher scores indicate greater levels of depressive symptoms.
Pain Catastrophizing as assessed by the Pain Catastrophizing Scale | Baseline - Final assessment (average 1 week post treatment)
  The Pain Catastrophizing Scale (PCS) is a 13 item survey assessing catastrophizing in context to pain. There are 13 items with 5-pt Likert responses.
  There are several subscales. Scoring Procedure: The PCS total score is computed by summing responses to all 13 items (0-52).
  Subscales:
  Rumination: Sum of items 8, 9, 10, 11 (0-16). Magnification: Sum of items 6, 7, 13 (0-12). Helplessness: Sum of items 1, 2, 3, 4, 5, 12 (0-24).
Pain-related fear of movement as assessed by the Tampa Scale Kinesiophobia | Baseline - Final assessment (average 1 week post treatment)
  The Tampa Scale Kinesiophobia (TSK) is a 17 item assessment of fear of movement. This uses a 5-pt Likert scale from 1 = Strongly Disagree to 4 = Strongly Agree.
  Scoring Procedure: Sum items Range: 17-68 Subscale Harm/Somatic Items: 3, 5, 6, 9, 11, 15 Subscale Avoidance Items: 1, 2, 7, 10, 13, 14, 17
Mood and Affect as assessed by the Positive and Negative Affect Scale | Baseline - Final assessment (average 1 week post treatment)
  The Positive and Negative Affect Scale (PANAS) measures mood of participants. This is a 20 item survey with 5 pt Likert response indicating to what degree the participant feels those emotions. There is a positive and negative subscale.
  Higher positive affect score indicates greater positive emotions; higher negative affect score indicates greater negative emotions.
  Range of Scores: 0-40
Immersive Tendencies | Baseline only
  Immersive Tendencies are assessed by the Immersive Tendencies Questionnaire (ITQ). This is an 18-item survey. Item responses use a 7 point Likert scale. Subscales include: focus, involvement, emotions, and play. Each subscale is scored by summing items. A total score is scored by summing all items.
  Range of total score: 18-126 Focus range of scores: 5-35 Involvement range of scores: 5-35 Emotions range of scores: 4-28 Play range of scores: 3-21 Higher scores indicate higher immersive tendencies overall and in each sub-scale.
Absorption Tendencies | Baseline Only
  Tellegen Absorption Scale is a 34-item multi-dimensional measure that assesses imaginative involvement and the tendency to become mentally absorbed in everyday activities. Item responses are on a 5-point Likert scale. Items are summed to score.
  Range of scores: 0-136. Higher scores indicate greater levels of absorption.
Video Game History | Baseline Only
  History of playing video games.
Patient Treatment Evaluation as assessed by the Modified Treatment Evaluation Inventory | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by Treatment Evaluation Inventory. This is a 9 item scale with a 5-point Likert responses for each question. The items are scored by summing all items.
  Range of scores: 9-45. A higher score indicates greater acceptance of treatment.
Patient Treatment Evaluation as assessed by Semi-structured Qualitative interviewing | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by semi-structured interviewing. Qualitative feedback from participant experience will be assessed by thematic analyses.
Daily intervention feedback questions | Baseline - Final assessment (average 1 week post treatment)
  The daily intervention feedback questions are 7 items that assess the individuals feelings and experiences during that daily intervention session.
  0-10 Likert scale
  Each item is it's own scale.
  Higher scores indicate more enjoyment/usefulness/demand/awareness/concern/mood.
Patient Treatment Evaluation as assessed by the Usefulness, Satisfaction, and Ease of Use Questionnaire | Final assessment (average 1 week post treatment)
  The Usefulness, Satisfaction, and Ease of Use Questionnaire (USE, Lund, 2001) measures the subjective usability of a product or service. It is a 30-item survey that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. This metric can be applied to various scenarios of usability assessment because it is non-proprietary and technology-agnostic. is a 30 item survey.
  Each item is presented on a 7-point Likert scale from strongly disagree = 1 to strongly agree. = 7
  Each subscale is calculated by averaging all items in subscale. Usefulness: items 1-8 Ease of use: items 9-19 Ease of Learning: items 20-23 Satisfaction: items 24-30
  Range of scores for each subscale: 1-7 Scoring Interpretation: Higher score indicates greater usefulness, satisfaction, and ease of use.
Patient Treatment Evaluation as assessed by the Patient Global Impression of Change Scale | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by the Patient Global Impression of Change. This is a one item 7 point Likert item assessing improvement of the participants overall status.
  Item responses:
  1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse
Video Game Preferences as assessed by the BrainHex | Final assessment (average 1 week post treatment)
  Video game preferences will be assessed by the BrainHex. The BrainHex provides a tool for designing gameplay and understanding motivations for play.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States